CLINICAL TRIAL: NCT03953859
Title: Investigation of Cellular DNA Repair Capacity in Human Preimplantation Embryos
Brief Title: Embryo DNA Repair Capacity Project
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-UK-01
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gamete donors: healthy male and female game donors to undergo routine gamete donation process
  Interventions: Genetic: double strand break
- Infertile Couple: Couples undergoing routine IVF to treat their infertility

INTERVENTIONS:
Genetic: double strand break — an induction of a double strand break will be made in the embryos generated for this research and the repair mechanism observed
  Groups: Gamete donors

SUMMARY:
The mail aim of the present study is to use molecular methods to analyze the ability of human preimplantation embryos to repair their DNA

DETAILED DESCRIPTION:
The main aim of the present study is to investigate the DNA repair pathways of preimplantation embryos, examining the events that take place following induction of a DSB at a unique targeted site. The investigators aim to address questions concerning the functionality of the DNA repair mechanism(s) in developing embryos, before and after genome activation.

ELIGIBILITY:
Inclusion Criteria:

* gamete donors: be at least 21 years of age, in good health and eligible to donate their games through the standard gamete donation programs
* IVF couples: any couples proceeding with a routine IVF cycle

Exclusion Criteria:

* less than 21 years of age
* inability to provide informed consent

Ages: 21 Years to 42 Years | Sex: All
Age Groups: Adult
Study Population: Healthy volunteer subjects will be recruiting from amongst the gamete donor population and patients undergoing in vitro fertilization (IVF) for treatment of their infertility
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
repair of double strand break in DNA | up to 12 days
  targeted deep sequencing to identify the presence of the double strand break in the DNA and subsequent repair ability of the embryo

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medicine Assoicates of New Jersey, Basking Ridge, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No